CLINICAL TRIAL: NCT06401603
Title: A Phase I Study of Decitabine, Lisaftoclax, and Olverembatinib in Patients With Advanced Chronic Myeloid Leukemia and Philadelphia Chromosome-Positive Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0032; NCI-2024-03867 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Advanced Chronic Myeloid Leukemia; Philadelphia Chromosome-Positive Acute Myeloid Leukemia
MeSH Terms: interventions — Decitabine; olverembatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Participants enrolled in Phase I, the dose of lisaftoclax you receive will depend on when a participants join this study. Up to 2 dose levels of lisaftoclax will be tested. Between 3-12 participants will be enrolled at each dose level.
  Interventions: Drug: Decitabine; Drug: Listaftoclax; Drug: Olverembatinib
- Phase 2 (Experimental): Participants enrolled in Phase II, participants will receive lisaftoclax at the recommended dose that was found in Phase I
  Interventions: Drug: Decitabine; Drug: Listaftoclax; Drug: Olverembatinib

INTERVENTIONS:
Drug: Decitabine — Given by IV
  Other Names: Dacogen
Drug: Listaftoclax — Given by PO
Drug: Olverembatinib — Given by PO

SUMMARY:
To find the recommended doses of lisaftoclax and olverembatinib that can be given in combination with decitabine to participants with advanced CML and Ph+ AML.

DETAILED DESCRIPTION:
Primary Objectives

• To establish the minimum safe and biologically-effective dose of lisaftoclax and olverembatinib in combination with decitabine

Secondary Objectives

* To determine the rate of conversion to CML-CP for participants with advanced phase CML or complete remission (CR)/CR with incomplete hematology recovery (CRi) for participants with Ph+ AML, within 4 cycles of combination therapy
* To assess other efficacy endpoints (CR rate, measurable residual disease negativity by flow cytometry, rates of CCyR, MMR, MR4 and MR4.5, relapse-free survival, overall survival)
* To assess proportion of participants proceeding to allogeneic hematopoietic stem cell transplantation
* To determine the safety of the combination regimen

Exploratory Objectives

* To evaluate the impact of olverembatinib monotherapy on signaling pathways and apoptotic protein expression
* To assess relationship between baseline signaling pathway activation and apoptotic protein expression on response and long-term outcomes such as overall survival (OS) and relapse free survival (RFS).

ELIGIBILITY:
Inclusion Criteria:

a) Diagnosis: Age ≥18 years with CML-AP, CML-MBP, or Ph+ AML by WHO 2016 criteria.

* Participants must have been intolerant or resistant to at least one prior BCR::ABL1 TKI

  2. Performance status ≤3 (ECOG Scale).

  3. Adequate liver, cardiac, renal and pancreatic function as defined by the following criteria:
  1. Total serum bilirubin < 1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome, hemolysis or the underlying leukemia approved by the PI
  2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 3 x ULN, unless due to the underlying leukemia approved by the PI
  3. Creatinine clearance ≥30 mL/min
  4. Serum amylase or lipase < 1.5 x ULN

     4. Ability to understand and the willingness to sign a written informed consent document

     5. Willingness to use adequate contraception prior to study entry, for the duration of study participation, and for 6 months after completion of study participation. For women of child-bearing potential, adequate methods of contraception include: complete abstinence,, hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device (IUD), tubal Ligation or hysterectomy, subject/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide.

     Exclusion Criteria:
     1. Participants who have previously received lisaftoclax or olverembatinib
     2. History of acute pancreatitis within 1 year of study or history of chronic pancreatitis
     3. Active grade III-V cardiac failure as defined by the New York Heart Association Criteria
     4. Clinically significant and uncontrolled cardiovascular disease, including but not restricted to:

        i. Myocardial infarction (MI), stroke, revascularization, unstable angina, or transient ischemic attack within 6 months.

        ii. Left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards prior to enrollment.

        iii. Diagnosed or suspected congenital long QT syndrome. iv. Clinically significant atrial or ventricular arrhythmias (such as uncontrolled, clinically significant atrial fibrillation, ventricular tachycardia, ventricular fibrillation, or Torsades de pointes) as determined by the treating physician.

        v. Prolonged QTc interval on pre-entry electrocardiogram (> 480 msec) unless corrected after electrolyte replacement.

        vi. History of venous thromboembolism including deep venous thrombosis or pulmonary embolism within the past 3 months, excluding line associated DVT of the upper extremity vii. Uncontrolled hypertension (diastolic blood pressure >100mmHg; and systolic >150mmHg).
     5. Active serious infection not controlled by oral or intravenous antibiotics (e.g. persistent fever or lack of improvement despite antimicrobial treatment).
     6. Active central nervous system leukemia
     7. Known human immunodeficiency virus (HIV) seropositive, unless well-controlled on stable doses of anti-retroviral therapy.
     8. Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection Note: Participants who have isolated positive hepatitis B core antibody (ie, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Participants who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.
     9. Participants with a prior or concurrent malignancy whose natural history or treatment is not anticipated to interfere with the safety or efficacy assessment of the investigational regimen may be included only after discussion with the PI
     10. Consumed strong inducer of CYP3A or p-glycoprotein within 14 days of study enrollment, or 5 half-lives, whichever is longer. Agents include but are not limited to: carbamazepine, phenytoin, rifampin, and St. John's wart
     11. Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator. Prior recent treatment with corticosteroids, hydroxyurea, cytarabine (up to 2 g/m2 given for cytoreduction within the preceding 7 days) and/or an FDA-approved BCR::ABL1 TKI is permitted.
     12. Inability to swallow
     13. Pregnant or breastfeeding women will not be eligible
     14. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Decitabine, Lisaftoclax, and Olverembatinib or other agents used in study.
     15. Participants with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Short, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org